CLINICAL TRIAL: NCT00535275
Title: Comparison of 2 Chemotherapy Regimens in Non-small-cell Lung Cancer (NSCLC) Patients Relapsing After Surgery and Peri-operative Chemotherapy. A Randomized Phase III Study.
Brief Title: NSCLC Relapse Therapy After Surgery and Peri-operative Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Final analysis done, follow-up of patients no more necessary
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0702
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC relapse after adjuvant chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Chemotherapy with platine
- B (Active Comparator): Docetaxel monotherapy
  Interventions: Drug: Chemotherapy without Cisplatine

INTERVENTIONS:
Drug: Chemotherapy with platine — Docetaxel 75 mg/m² D1 + Cisplatine 75 mg/m² or Carboplatin AUC5 D1 (D1=D22, 4 cycles) Docetaxel 75 mg/m² D1 (D1=D22, 2 cycles if disease control)
  Arms: A
Drug: Chemotherapy without Cisplatine — Docetaxel 75 mg/m² D1 (D1=D22, 4 cycles) Docetaxel 75 mg/m² D1 (D1=D22, 2 cycles if disease control)
  Arms: B

SUMMARY:
Relapses after perioperative chemotherapy and surgery

DETAILED DESCRIPTION:
As chemotherapy gains wider acceptance for the treatment of earlier stages of NSCLC, particularly in the adjuvant and neoadjuvant setting, physicians face a growing population of high performance status patients who have relapsed after their first-line chemotherapy. The type of second-line chemotherapy after initial adjuvant or neoadjuvant treatment with a platinum-based regimen remains largely undefined. Some might consider rechallenging patients with a platinum based doublet whereas others might treat these patients with a monochemotherapy (pemetrexed or docetaxel).

Most relapses occurring after perioperative chemotherapy and surgery are non surgical locally advanced relapses or metastatic diseases.

Some differences exist between these post surgical relapses and the progressions occurring after the first line non surgical treatment of a stage III/IV.

* Patients are most often in a good condition (performance status 0-1).
* Progression is often asymptomatic and diagnosed in the post surgical follow up.
* The dose of chemotherapy previously administered is lower than that administered in first line of a stage III/IV.
* The time between the first line of treatment and the treatment of the relapse is longer.

These differences might be associated with a more chemosensitive disease and thus might be the rationale of using a platinum containing doublet instead of the classical mono chemotherapy docetaxel or pemetrexed.

Thus, the current study has been designed to answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed inoperable non-small cell-lung cancer not eligible for curative radio-therapy (local or metastatic relapse).
* Previous history of adjuvant or neoadjuvant chemotherapy (at least 2 full cycles of a platinum containing regimen)
* Initial stage pT1N0 to pT3N2 (TNM classification 1999), complete resection. T4 tumours (several nodules in the same lobe) and M1 tumours (several nodules in the same lung) N0-2 completely resected are allowed to inclusion. Histological complete response tumours (pT0N0) after neoadjuvant chemotherapy are allowed to inclusion.
* At least one unidimensionally measurable disease (RECIST criteria) (lesions must have clearly defined margins on X-ray, CT-scan, MRI or ultra-sound (US) examination and should measure at least 1 cm if assessed by CT, MRI or US and at least 2 cm if assessed by X-ray, target lesions should be selected outside a previously irradiated field ). PET scans and ultra sonography are not allowed
* ECOG Performance status 0 to 1).
* Patients with adequate biological functions:
* Written informed consent from patient.
* The effects of docetaxel, cisplatin and carboplatin on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because docetaxel, cisplatin and carboplatin as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Life expectancy > 12 weeks
* Patient compliance and geographic proximity that allow adequate follow-up.
* Patient affiliated to a social insurance program

Exclusion Criteria:

* Previous treatment with docetaxel.
* Hypersensitivity to docetaxel, cisplatin, carboplatin or polysorbate 80 (excipient).
* Previous history of cancer other than Non small cell lung cancer, in situ carcinoma of the uterine cervix and basal cell carcinoma of the skin.
* Patients previously treated by an investigational agent in the last 30 days.
* Patient treated with preoperative platin based chemotherapy, achieving a progression of disease after treatment evaluation.
* Patients non responders to preoperative chemotherapy and whose tumor specimen did not disclose any necrosis nor tumoral modification thus confirming the lack of chemosensitivity to platin based chemotherapy
* Patient treated with platin based adjuvant chemotherapy, relapsing within the first 6 months after surgery.
* Patients with a peripheral neuropathy grade CTC >= 2
* Patients unable to fulfill protocol requirements
* Serious concomitant morbidity incompatible with the study (at the discretion of the investigator).
* Relapse within the month following lung cancer resection or adjuvant chemotherapy
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Significant loss of weight (> 10 %) in the 6 weeks preceding patient selection.
* Concomitant administration of another anti cancer treatment
* Pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued.
* Patient under legal protection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Denis Moro-Sibilot, Pr, Principal Investigator — University Hospital, Grenoble
Locations (78):
- France (78):
  - Centre Hospitalier, Aix-en-Provence
  - Annemasse - CH, Ambilly
  - Annecy - CH, Annecy
  - Auxerre - Polyclinique, Auxerre
  - Auxerre - CH, Auxerre
  - CH de la Côte Basque, Bayonne
  - Beauvais - CH, Beauvais
  - CHU Besancon - Pneumologie, Besançon
  - Blois - CH, Blois
  - APHP - CHU Avicenne - Oncologie Medicale, Bobigny
  - Boulogne - Ambroise Paré, Boulogne
  - Caen - Centre François Baclesse, Caen
  - CHU - Pneumologie, Caen
  - Calais - CH, Calais
  - CH de Cannes, Cannes
  - Chambray Les Tours - Clinique Léonard de Vinci, Chambray-lès-Tours
  - Chauny - CH, Chauny
  - Chevilly-Larue - CH, Chevilly-Larue
  - Hôpital de Cholet - Pneumologie, Cholet
  - Hôpital Percy-Armées - Pneumologie, Clamart
  - Hôpitral Gabriel Montpied - Pneumologie, Clermont-Ferrand
  - CH, Colmar
  - CHI Créteil, Créteil
  - Dax - CH, Dax
  - Dijon - CHU, Dijon
  - Epinal - CH, Épinal
  - CHU, Grenoble
  - Saint Omer - CHI, Helfaut
  - La Roche Sur Yon - CH, La Roche-sur-Yon
  - Chartres - CH, Le Coudray
  - Le Mans - Centre Hospitalier, Le Mans
  - Limoges - Hôpital du Cluzeau, Limoges
  - CH de Longjumeau, Longjumeau
  - HCL - Croix-Rousse, Lyon
  - Lyon - Clinique Mutualiste, Lyon
  - Hôpital Louis Pradel, Lyon
  - Hôpital Nord - Oncologie Multidisciplinaire & Innovations Thérapeutiques, Marseille
  - Maubeuge - Polyclinique du Parc, Maubeuge
  - CH de Macon, Mâcon
  - Meaux - CH, Meaux
  - Mont de Marsan - CH, Mont-de-Marsan
  - Centre Hospitalier, Montélimar
  - Moulins - CH, Moulins
  - Mulhouse - CH, Mulhouse
  - CHU, Nancy
  - Nanterre - CH, Nanterre
  - Nantes - Centre René Gauducheau, Nantes
  - CH Nevers, Nevers
  - Nîmes - Clinique Valdegour, Nîmes
  - Orléans - CH, Orléans
  - APHP - Hopital Tenon - Pneumologie, Paris
  - GH Paris Saint-Joseph, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Catalan d'Onologie, Perpignan
  - Perpignan - Ch, Perpignan
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - Centre Hospitalier, Rambouillet
  - Reims - CHU, Reims
  - Institut Jean Godinot, Reims
  - Rodez - CH, Rodez
  - Roncq - Clinique Saint-Roch, Roncq
  - Roubaix - CH, Roubaix
  - CH de Saint-Brieuc, Saint-Brieuc
  - Saint Nazaire - Centre Etienne Dolet, Saint-Nazaire
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Saint Quentin - CH, Saint-Quentin
  - Saint-Malo - CH, St-Malo
  - CHU Lyautey - Pneumologie, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpitaux du Léman - Pneumologie et Maladies Infectieuruses, Thonon-les-Bains
  - Toulon - CHI, Toulon
  - Toulouse - CHU Larrey, Toulouse
  - Tours - CHU, Tours
  - Troyes - CH, Troyes
  - Valenciennes - Clinique, Valenciennes
  - CHI de la Haute-Saône - Pneumologie, Vesoul
  - Vienne - CH, Vienne
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- See also: IFCT official website — http://www.ifct.fr